CLINICAL TRIAL: NCT00330096
Title: Effects of Hesperidin on Bone Mineral Density and Bone Metabolism of Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Centre de Recherche en Nutrition Humaine. Clermont-Ferrand, France (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05.12NRC
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Osteoporosis, Osteopenia
Keywords: bone loss, osteoporosis, prevention, hesperidin
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Hesperidin

ARMS (2):
- Hesperidin-rich food (Experimental)
  Interventions: Drug: Hesperidin
- No intervention: Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hesperidin
  Arms: Hesperidin-rich food
Other: Placebo
  Arms: No intervention: Placebo

SUMMARY:
Fruits and vegetables are rich in a variety of flavonoids with antioxidant properties. These compounds may be partially responsible for some of the positive links found between fruits and vegetables intake and higher bone mineral density in adults and children. Several animal studies have shown that consumption of onions (which are rich in quercetin), rutin (a quercetin glycoside) and resvatrol (found in red wine) inhibits ovariectomy induced bone loss in rats. One of the most studied flavonoids with respect to bone health is the soy isoflavones. However, consumption of soy products is relatively low in Western countries. One the other hand, a flavonoid such as hesperidin, found mostly in oranges is much more abundant in the Western diet. Citrus juice consumption has been demonstrated to prevent bone loss in male orchidectomized rats while specifically feeding hesperidin has been shown to prevent bone loss in ovariectomized mice and rats. However, to date no clinical prove has been obtained for these benefits.Therefore the aim of this study is to investigate the effect of hesperidin in preventing bone loss in postmenopausal women. This study is designed as a 2-year, double blind, placebo-controlled, two arm, and parallel group study. The primary outcome measure is change in bone mineral density (BMD) while the secondary outcome measures are changes in bone resorption and formation markers as well as body composition. The women are randomised to consume 2 servings of hesperidin-rich food or food without hesperidin but with the same taste & appearance (placebo). Subjects will undergo medical screening, anthropometry, physical activity, dietary assessments and BMD before randomisation into placebo or active group. Follow-up measurements are made at 3-month intervals (for blood and urine collection) and 6-month intervals for bone mineral density. Side effects are also being monitored during each visit.

ELIGIBILITY:
Inclusion Criteria:

50 - 65 years, Caucasian female Community dwelling women· Within 3-10 years post-menopause (natural or surgical) and FSH > 20UI/L· Generally healthy as determined by standard medical assessment on physical and mental health · Normal weight as determined by BMI (19≤ BMI ≤29)· Affiliated to National Health Insurance (Sécurité Sociale)· Willing to comply with the study procedures· Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data· Having received both oral and written explanations about the study· Having provided her written informed consent

Exclusion Criteria:

·Intestinal or severe metabolic diseases / disorders such as diabetes, renal, hepatic or pancreatic diseases / disorders, ulcer, hyperthyroidism, malignancy, chronic malnutrition· Have had major gastrointestinal surgery· Osteoporosis (defined by T-score of £ -2.5 SD at hip and/or spine)· Very low BMD at hip and "and/or" spine, indicating high risk of osteoporosis (T-score £ -2.0 SD)· Severe scoliosis that could interfere with BMD measurements· On therapy with drugs known to interfere with bone metabolism such as steroids, vitamin D or its derivatives, bisphosphonates, strontium ranelate, PTH, calcitonin, raloxifene, etc. · On hormone replacement therapy (HRT) previous 3 months before entering the study Taking medications containing hesperidin (e.g.Daflon) or known to interfere with hesperidin (statins, therapy for circulatory disorders, anti-depressants)Known to have allergic reactions to citrus-containing foods· Taking regular calcium (> 500 mg/day) and vitamin D (> 400 IU/day) supplements Hypercholesterolemia with HDL < 1,30 mmol/L (0,5 g/L)· Having a baseline calcium intake of below 800 mg/day and 25-OH vitamin D status of below 25 nmol/L or above 200 nmol/L· Have an alcohol intake > 2 glasses of wine per day (3dL/day), or > 2 beers (3dL/d) or > 1 shot glass of hard alcohol· Heavy smoker (more than 10 cigs a day) and for pipe/cigars· Blood donation less than 3 months before the beginning of the study· Currently participating or having participated in another clinical trial during past 1 year prior to the beginning of this study, this depending on the type of previous study· Special dietary habits (vegetarians)· Phytoestrogens or antioxidants (dietary supplements) consumption· Physical activity > 10 hours / week

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2006-03; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Bone mineral density

SECONDARY OUTCOMES:
Serum markers of bone resorption and bone formationChanges in body composition

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noelle Horcajada, PhD, Principal Investigator — INRA de Theix Laboratoire des Maladies Métaboliques et Micronutriments
Locations (1):
- Centre de Recherche en Nutrition Humaine. Laboratoire de Nutrition Humaine, Clermont-Ferrand, Auvergne, France